CLINICAL TRIAL: NCT06427733
Title: Green Banana Peel Extract for Stasis Dermatitis Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sponsor
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Stasis Dermatitis
Keywords: Stasis dermatitis; Hyperpigmentation; banana skin; Musa sapientum
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group without green banana peel (Placebo Comparator): SPF 30 and Placebo Control Group will use SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract
  Interventions: Biological: Placebo comparator
- Study Group with green banana peel (Active Comparator): SPF 30 and pharmaceutical formulation with green banana peel In Study Group, in addition to the SPF 30 sunscreen, a pharmaceutical formulation containing the extract of the green banana peel will be used.
  Interventions: Biological: Active Comparator

INTERVENTIONS:
Biological: Placebo comparator — SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract Control Group will use SPF 30 sunscreen plus pharmaceutical formulation without green banana peel extract
  Arms: Control Group without green banana peel
Biological: Active Comparator — SPF 30 sunscreen and pharmaceutical formulation containing green banana peel extract
  Arms: Study Group with green banana peel

SUMMARY:
To develop and evaluate a pharmaceutical formula based on green banana peel extract for the treatment of stasis dermatitis.

DETAILED DESCRIPTION:
Objective: to develop and evaluate a pharmaceutical formula based on green banana peel extract for the treatment of stasis dermatitis. Methods: it will be a clinical, interventional, longitudinal study, random sampling, Sample will have 20 patients divided into two groups. In the Control Group, a moisturizing cream with SPF 30 sunscreen plus a pharmaceutical formulation without green banana peel extract will be used, and in the Study Group, in addition to the SPF 30 sunscreen, a pharmaceutical formulation containing green banana peel extract will be used. Patients will undergo treatment for 90 days, applying the formulation twice a day, evaluated every 45 days through clinical, photographic and Chromatic Palette evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stasis dermatitis.
* Patients aged 18 years or over and 60 years or less.
* Patients who agree to participate in the study. -

Exclusion Criteria:

* Patients who have other types of hyperchromia in the legs.
* Patients known to have an allergic reaction to bananas.
* Patients who give up, for any reason, to continue treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Occurence of stasis dermatitis | 3 months
  Macroscopic Analysis: The occurrence of stasis dermatitis will be determined by hyperpigmentation, measured using the Chromatic Palette. Changes in skin color vary from ecchymosis, hematomas, erythema, hyperpigmentation, hypochromia and cyanosis. The focus of our study being hyperpigmentation, the shades vary between brownish, grayish and reddish, depending on the evolution, clinical duration and skin color and severity of stasis dermatitis. The positioning of colors on a gradient scale in columns and lines favors the comparative process and location between nearby shades corresponding to the observed evidence. The inclusion of codes makes it possible to locate and classify skin colors in the situations in which they will be evaluated. In the final version that will be used, there are 72 color possibilities.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R dos Anjos Mendonça, PhD, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Vale do Sapucaí University, Pouso Alegre, Minas Gerais, Brazil